CLINICAL TRIAL: NCT06970249
Title: The Differences Between the Effects of Intraoperative vs Postoperative Preferred Music on Emergence Agitation or Delirium in Elderly Patients: A Prospective Randomized Controlled Trial
Brief Title: Music Timing for Emergence Delirium in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Wonkwang UH18
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Delirium on Emergence; Elderly; Satisfaction, Patient
MeSH Terms: conditions — Emergence Delirium; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Patient-preferred music (e.g., classical, jazz, ambient) will be selected preoperatively from a standardized list and delivered via headphones at 40-60 dB, verified by a sound meter.
  1. Intraoperative music will be played from induction to extubation;
  2. Postoperative music will be provided for 60 minutes following extubation in the PACU.
  3. The control group will receive standard care with ambient sounds.
Who Masked: Outcomes Assessor
Masking Description: "Outcome assessors (PACU nurses) will be blinded to group allocation. Participants, care providers, and investigators will not be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group received standard care with ambient sounds.
- Intraoperative (Active Comparator): Patient-preferred music (e.g., classical, jazz, ambient) will be selected preoperatively from a standardized list and delivered via headphones at 40-60 dB, will be verified by a sound meter. Intraoperative music will run from induction to extubation
  Interventions: Behavioral: Music intervention
- Postoperative (Active Comparator): Patient-preferred music (e.g., classical, jazz, ambient) will be selected preoperatively from a standardized list and delivered via headphones at 40-60 dB, will be verified by a sound meter. Postoperative music will be provided for 60 minutes after extubation in the PACU.
  Interventions: Behavioral: Music intervention

INTERVENTIONS:
Behavioral: Music intervention — Patient-preferred music (e.g., classical, jazz, ambient) will be selected preoperatively from a standardized list and delivered via headphones at 40-60 dB, verified by a sound meter.
  Arms: Intraoperative; Postoperative

SUMMARY:
Emergence delirium (ED) after general anesthesia prolongs recovery, increases complications, and adds to nursing workload in elderly patients. Although music has been shown to alleviate anxiety and agitation, the optimal timing for its delivery and the factors that predict its effectiveness remain unclear.

This trial will compare preferred music played during surgery versus music played after surgery to see how each affects the incidence, the severity, and the duration of ED in older adults, and to identify which patient characteristics predict ED.

DETAILED DESCRIPTION:
Study Design and Participants This prospective, single-blind, randomized controlled trial will be conducted following approval by the Institutional Review Board of Wonkwang University Hospital (IRB No. [2025-04-021-0045]). Written informed consent will be obtained from all participants. The study will adhere to the 2013 Declaration of Helsinki.

The investigators will enroll adults aged 65 years or older with American Society of Anesthesiologists (ASA) physical status I-III scheduled for elective surgery lasting 1-3 hours under general anesthesia. All participants will have a Mini-Mental State Examination (MMSE) score of 20 or higher and no significant hearing impairment. Patients undergoing emergency procedures, those with severe psychiatric illness, an MMSE score below 20, or any condition preventing informed consent will be excluded.

Randomization and Blinding A computer-generated random sequence will be created using Stata 17.0 (StataCorp, College Station, TX, USA), employing block randomization stratified by age group (65-75 vs. >75 years), sex, and surgery type. Allocation to one of three groups-intraoperative music, postoperative music, or control-will be concealed in sealed, opaque envelopes. PACU nurses assessing outcomes will remain blinded; anesthesiologists and PACU staff administering music interventions will not participate in data collection.

Interventions General anesthesia will be induced with propofol (2 mg/kg), maintained with sevoflurane (BIS 40-60), and supplemented with remifentanil (0.05-0.2 µg/kg/min). No benzodiazepine premedication will be administered. Patient-preferred music (e.g., classical, jazz, ambient) will be selected preoperatively from a standardized list and delivered via headphones at 40-60 dB, verified by a sound meter. Intraoperative music will be played from induction to extubation; postoperative music will be provided for 60 minutes following extubation in the PACU. The control group will receive standard care with ambient sounds. Intraoperative hypotension (mean arterial pressure <20% of baseline) will be treated with ephedrine (5-10 mg), and postoperative pain will be managed with fentanyl (0.5 µg/kg) as needed.

Outcome Measures The primary outcome will be the incidence of ED, defined as a Richmond Agitation-Sedation Scale (RASS) score ≥+1 within 60 minutes after extubation, assessed every 15 minutes by two trained PACU nurses (expected inter-rater κ = 0.85). Secondary outcomes will include severity of ED (highest RASS score within 60 minutes), duration of ED (minutes from extubation to RASS ≤ 0), postoperative pain (VAS, 0-10, assessed every 15 minutes for 60 minutes), patient satisfaction (5-point Likert scale, 1 = very dissatisfied, 5 = very satisfied, at PACU discharge), adverse events (including incidence of nausea, vomiting, respiratory depression, and other complications), and preoperative anxiety.

Preoperative anxiety will be measured using the State-Trait Anxiety Inventory (STAI-S); scores range from 20 to 80, with higher scores indicating greater anxiety (including 10 reverse-scored items). All data will be recorded using a standardative outcomes.ized Case Report Form, encompassing demographic information, MMSE scores, anesthetic details, and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have a Mini-Mental State Examination (MMSE) score of 20 or higher and no significant hearing impairment.

Exclusion Criteria:

* Investigators will exclude patients undergoing emergency procedures, those with severe psychiatric illness, MMSE below 20, or any condition preventing informed consent.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
the incidence of emergence delirium (ED) | will be assessed every 15 minutes and during staying in the Postanesthesia care unit (PACU)
  wil be defined as a Richmond Agitation-Sedation Scale (RASS) score ≥+1 within 60 minutes after extubation.

SECONDARY OUTCOMES:
The severity of emrgence delirium (ED) | within 60 minutes in the PACU
  highest RASS score
The duration of ED | within 60 minutes in the PACU
  minutes from extubation to RASS ≤ 0
Postoperative pain | will be assessed every 15 minutes and during staying in the Postanesthesia care unit (PACU)
  visual analogue scale (VAS, 0-10)
Patients satisfaction | When patients leave from PACU.
  5-point Likert scale, 1 = very dissatisfied, 5 = very satisfied,
preoperative anxiety | the day before the operation
  the State-Trait Anxiety Inventory (STAI-S, 20-80, with 10 positively worded items reverse-scored).

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwag UH, Iksan, Jeollabukdo, South Korea

IPD SHARING:
Plan to Share IPD: No
The data are available from the corresponding author upon reasonable request, subject to institutional approval.

REFERENCES:
- [Result] Golubovic J, Neerland BE, Aune D, Baker FA. Music Interventions and Delirium in Adults: A Systematic Literature Review and Meta-Analysis. Brain Sci. 2022 Apr 28;12(5):568. doi: 10.3390/brainsci12050568. PMID 35624955